CLINICAL TRIAL: NCT02473419
Title: Neurobiological Basis of Response to Vayarin in Adults With ADHD: an fMRI Study of Brain Activation Pre and Post Treatment
Acronym: VAYA-fMRI
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: New York University (Other); Enzymotec (Industry); The Medical Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 15-0399
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: ADHD
Keywords: Medical food; ADHD; Vayarin; Fish Oil
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Vayarin: Vayarin x 16 weeks
  Interventions: Drug: Vayarin
- Placebo: Placebo x 16 weeks
  Interventions: Drug: Placebo
- Vayarin and Placebo: Placebo x 8 weeks and then Vayarin x 8 weeks
  Interventions: Drug: Vayarin; Drug: Placebo

INTERVENTIONS:
Drug: Vayarin
  Groups: Vayarin; Vayarin and Placebo
Drug: Placebo
  Groups: Placebo; Vayarin and Placebo

SUMMARY:
The objective of this research is to use functional magnetic resonance imaging (fMRI) with a neuropsychological task to test the prefrontal mechanism of action of the medical food Vayarin.

DETAILED DESCRIPTION:
The investigators prior research suggests that effective non-stimulant treatments for ADHD act through key prefrontal regions that subserve inhibitory and executive functions, although different medications may achieve these effects via distinct mechanisms. The objective of this research is to use functional magnetic resonance imaging (fMRI) with a face go/no-go task to test the prefrontal mechanism of action of the medical food Vayarin. Participants are not treated at the Icahn School of Medicine, but instead will be recruited from trials of Vayarin that are enrolling and treating participants at New York University and The Medical Research Network.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible to enroll in the Vayarin clinical study according to screening visit will be asked to participate in the fMRI study.
* Must be willing and able to perform fMRI scanning
* Must maintain compliance to their trials' protocols

Exclusion Criteria:

* pre-existing medical or psychological condition that precludes scanning (e.g., claustrophobia, morbid obesity)
* implanted medical device (e.g., pacemaker)
* metal in the body that cannot be removed (e.g., braces)
* pregnancy
* concomitant use of anti-hypertensives or any other medications affecting the blood oxygenation level-dependent (BOLD) signal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be subjects participating in a Vayarin clinical trial being conducted at NYU and The Medical Research Network in NYC.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2015-05; Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Change in the emotional go/no-go task | Baseline and 16 weeks
  Change in the emotional go/no-go task performed in the fMRI scanner at 16 weeks as compared to baseline

SECONDARY OUTCOMES:
Change in the resting state fMRI | Baseline and 16 weeks
  Change in the resting state fMRI at 16 weeks as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Newcorn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States